CLINICAL TRIAL: NCT01866865
Title: Adaptation to Living With a BRCA l/2 Mutation in Carriers and Their Partners
Brief Title: Adaptation to Living With a BRCA1/2 Mutation
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913134; 13-HG-N134
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-11-22

CONDITIONS: Cancer Genetics
Keywords: BRCA1; BRCA2

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Background:

- Women who have a BRCA1/2 gene mutation have a very high risk of developing breast or ovarian cancer. They are also at increased risk of other developing other cancers. Male carriers are at increased risk for breast, prostate and other cancers. Testing for this mutation and living with this increased risk can be a source of stress for both people with the mutation and their partners. Researchers want to look at how well people adapt to living with this type of cancer risk over time.

Objectives:

- To see how women with the BRCA1/2 gene mutation and their partners adapt to the stress of long-term cancer risk.

Eligibility:

- Women at least 18 years of age who have a BRCA1/2 mutation, and their male or female partners.

Design:

* This study involves a one-time self-administered questionnaire. Participants will be recruited from local and national hereditary cancer support groups and cancer centers.
* There are two versions of the survey. One is for the woman with the BRCA1/2 gene mutation. The other is for her partner.
* The survey will ask about risk perception, cancer worry, risk-related stress, and coping and adaptation methods.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
The proposed study aims to describe adaptation and dyadic adjustment in unaffected BRCA1/2 carriers and their partners. It is not fully understood how women and their partners adapt to highrisk status over time, nor how different aspects of living at risk relate to this process. Neither psychological adaptation nor dyadic adjustment has been systematically measured in this population. This study is informed by Lazarus & Folkman s Transactional Model of Stress and Coping and modifications made to this model for use in studying dyadic relationships. A crosssectional research design will quantitatively explore the relationships between the appraisals and timing of risk-related stressors, dyadic coping, and the outcomes of adaptation and dyadic adjustment. Participants will be recruited from hereditary breast and ovarian cancer (HBOC) support groups, website postings, listservs, and clinic patient lists. They will have the option of completing either a paper or online version of the survey.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Participants will be women aged 18 or older who have a BRCA1/2 mutation and their (male or female) partners. Carriers must have no personal history of cancer, but partners will not be excluded based on cancer history. Participants will be asked to disclose their mutation status (BRCA1 or BRCA2), but no screening evaluation will be required. If only one member of a couple completes the survey, their data will be included in the individual level analysis, but excluded from the dyadic level analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2013-05-02; Primary Completion 2014-02-20 (Actual); Study Completion 2014-02-20 (Actual)

PRIMARY OUTCOMES:
the primary outcome is psychological adaptation | 1 time survey

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Berg CA, Upchurch R. A developmental-contextual model of couples coping with chronic illness across the adult life span. Psychol Bull. 2007 Nov;133(6):920-54. doi: 10.1037/0033-2909.133.6.920. PMID 17967089